CLINICAL TRIAL: NCT05960227
Title: Effect of Intravenous Iron Repletion on Renal Function in Patients With Iron Deficiency and Acute Kidney Injury, Clinical Trial
Brief Title: Effect of Intravenous Iron Repletion on Renal Function in Patients With Iron Deficiency and Acute Kidney Injury
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital Civil de Guadalajara (Other)
Responsible Party: Principal Investigator, Jonathan Samuel Chavez Iñiguez, Head of nephrology Jonathan Samuel Chavez Iñiguez MD., Hospital Civil de Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HCG
Record Dates: First submitted 2022-09-19; First posted 2023-07-25 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Anemia, Iron Deficiency; Acute Kidney Injury
Keywords: Acute kidney injury; Anemia; Iron deficiency
MeSH Terms: conditions — Anemia, Iron-Deficiency; Acute Kidney Injury; Anemia; Iron Deficiencies | interventions — Iron-Dextran Complex

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled clinical trial, method of randomization in blocks of 5 by frequency of occurrence. In patients with acute renal injury, patients will be allearorized to receive intravenous iron dextran in 1 single exhibition according to the Mg granted by the Virizzi formula compared to placebo.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Iron dextran IV (Experimental): In patients with acute renal damage, they will be aleatorized to receive the administration of intravenous iron dextran 1200mg in 1 single exhibition compared to placebo.
  Interventions: Drug: Iron dextran
- Placebo (Placebo Comparator): In patients with acute renal damage, they will be aleatorized to receive the administration of placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Iron dextran — Administration of 1.2g of iron dextran in infusion bolus as a loading strategy.
  Arms: Iron dextran IV
Drug: Placebo — 250ml of saline 0,9% for 4 hours insusion.
  Arms: Placebo

SUMMARY:
This clinical trial aims to carry out research on the effect on hemoglobin and renal function of intravenous administration of iron dextran as a repletion strategy in patients with iron deficiency anemia and acute kidney injury, in which the patient may benefit from this drug as it is expected to correct anemia, ferropenia and renal function parameters, when compared with a control group (placebo), the safety of the drug will also be assessed by recording adverse effects.

The investigators will point out with the patient the risks and benefits of their inclusion in this type of study and the investigators will attend to all the doubts that are generated, as well as immediately report to the research ethics committee any serious adverse effects. The results will be presented at national and international conferences and will be published in high-impact journals, and will also be the subject of a thesis to achieve the title of specialist.

DETAILED DESCRIPTION:
Acute kidney injury is a complication that occurs in up to 30% of hospitalized patients, iron deficiency has a high incidence in the critically ill patient population and has been associated with multiple complications such as the development of anemia and renal dysfunction. The presence of iron deficiency, anemia and acute kidney damage is a common combination in critically ill patients and it has been seen that iron deficiency promotes mitochondrial dysfunction and this can be improved with the correction of intravenous iron, as has happened in clinical trials of patients with acute heart failure, improving their clinical evolution.

There is insufficient evidence for the implementation of intravenous iron with the aim of improving the parameters of iron deficiency anaemia in patients with acute kidney injury.

To the knowledge of the investigators, there is no clinical trial that has explored this outcomes.

Primary objective:

• Renal function estimated in GFR at 3 months after randomization. Which will be evaluated by the estimation of the GFR by the equation CKD-EPI by serum creatinine

Secondary objectives: all of the following will be at hospital discharge and 28 days after hospital discharge between the intervention group (iron replacement) compared to the control group (placebo).

* ferritin value, (pg/dL)
* transferrin saturation (%)
* Hemoglobin (g/dL)
* serum creatinine (mg/dL)
* initiation of renal support therapy (any type of renal support such as: intermittent haemodialysis, peritoneal dialysis or continuous therapies)
* recovery of renal function, seen as decreased serum creatinine and approaching <0.3mg/dL of baseline creatinine
* death

Exploratory objectives:

• safety of intravenous iron administration compared to placebo: assessed for the occurrence of adverse events such as allergic reaction, hypotension, dyspnea, rash, erythema. These will be evaluated during the administration of the drug and during hospitalization frequently every 24 hours by the nephrology staff that includes the study researchers.

Our hypothesis is that intravenous iron dextran repletion during the treatment of acute kidney injury will improve the parameters of renal function, iron deficiency, anemia and also that it will be safe compared to placebo.

STUDY DESIGN Randomized, placebo-controlled clinical trial, method of randomization in blocks of 5 by frequency of occurrence. In patients with acute renal injury, they will be aleatorized to receive the administration of intravenous iron dextran in 1 single exhibition according to the Mg granted by the Virizzi formula compared to placebo.

The sample size determined 55 patients per group, with a standard deviation of 1.5.

The randomization process was carried out with the NCI Clinical Trial Randomization Tool:

https://ctrandomization.cancer.gov/

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients with acute kidney injury
* iron levels <13 μmol/L or a transferrin saturation <20%

Exclusion Criteria:

* AKI within the past three months
* less than 18 years old
* Chronic Kidney Disease grade 5
* chronic dialysis
* kidney transplant
* hospital stay less tahn 48 hours
* received any red blood cell transfusion before randomization
* missing data that would render analysis incomplete.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2023-01-06 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Renal function estimated in GFR at 3 months of randomization. Which will be evaluated by the estimation of the GFR by the equation CKD-EPI by serum creatinine. | 3 months of randomization
  The CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration) equation was developed in an effort to create a more precise formula to estimate glomerular filtrate rate (GFR) from serum creatinine and other readily available clinical parameters, especially at when actual GFR is >60 mL/min per 1.73m2.

SECONDARY OUTCOMES:
All of the following will be at hospital discharge and 28 days after hospital discharge between the intervention group (iron replacement) compared to the control group (placebo). | 28 days of discharge from hospital between iron dextran group and placebo group
  Ferritin value, (pg/dL)
Need of renal replacement therapy | 28 days of discharge from hospital between iron dextran group and placebo group
  Number of Participants with initiation of renal replacement therapy (any type of renal support such as: intermittent haemodialysis, peritoneal dialysis or continuous therapies)

OTHER OUTCOMES:
safety of intravenous iron | 1 day
  Number of Participants with adverse events such as allergic reaction, hypotension, dyspnea, rash, erythema. These will be evaluated during the administration of the drug and during hospitalization frequently every 24 hours by the nephrology staff that includes the study researchers.

CONTACTS AND LOCATIONS:
Locations (2):
- Mexico (2):
  - Hospital Civil de Guadalajara, Guadalajara, Jalisco
  - Jonathan Samuel Chávez Iñiguez, Guadalajara, Jalisco

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lameire NH, Bagga A, Cruz D, De Maeseneer J, Endre Z, Kellum JA, Liu KD, Mehta RL, Pannu N, Van Biesen W, Vanholder R. Acute kidney injury: an increasing global concern. Lancet. 2013 Jul 13;382(9887):170-9. doi: 10.1016/S0140-6736(13)60647-9. Epub 2013 May 31. PMID 23727171
- [Background] Siew ED, Davenport A. The growth of acute kidney injury: a rising tide or just closer attention to detail? Kidney Int. 2015 Jan;87(1):46-61. doi: 10.1038/ki.2014.293. Epub 2014 Sep 17. PMID 25229340
- [Background] Murugan R, Karajala-Subramanyam V, Lee M, Yende S, Kong L, Carter M, Angus DC, Kellum JA; Genetic and Inflammatory Markers of Sepsis (GenIMS) Investigators. Acute kidney injury in non-severe pneumonia is associated with an increased immune response and lower survival. Kidney Int. 2010 Mar;77(6):527-35. doi: 10.1038/ki.2009.502. Epub 2009 Dec 23. PMID 20032961
- [Background] Nisula S, Kaukonen KM, Vaara ST, Korhonen AM, Poukkanen M, Karlsson S, Haapio M, Inkinen O, Parviainen I, Suojaranta-Ylinen R, Laurila JJ, Tenhunen J, Reinikainen M, Ala-Kokko T, Ruokonen E, Kuitunen A, Pettila V; FINNAKI Study Group. Incidence, risk factors and 90-day mortality of patients with acute kidney injury in Finnish intensive care units: the FINNAKI study. Intensive Care Med. 2013 Mar;39(3):420-8. doi: 10.1007/s00134-012-2796-5. Epub 2013 Jan 5. PMID 23291734
- [Background] Bagshaw SM, George C, Dinu I, Bellomo R. A multi-centre evaluation of the RIFLE criteria for early acute kidney injury in critically ill patients. Nephrol Dial Transplant. 2008 Apr;23(4):1203-10. doi: 10.1093/ndt/gfm744. Epub 2007 Oct 25. PMID 17962378
- [Background] Ostermann M, Chang RW. Acute kidney injury in the intensive care unit according to RIFLE. Crit Care Med. 2007 Aug;35(8):1837-43; quiz 1852. doi: 10.1097/01.CCM.0000277041.13090.0A. PMID 17581483
- [Background] Hoste EA, Clermont G, Kersten A, Venkataraman R, Angus DC, De Bacquer D, Kellum JA. RIFLE criteria for acute kidney injury are associated with hospital mortality in critically ill patients: a cohort analysis. Crit Care. 2006;10(3):R73. doi: 10.1186/cc4915. Epub 2006 May 12. PMID 16696865
- [Background] Hoste EA, Bagshaw SM, Bellomo R, Cely CM, Colman R, Cruz DN, Edipidis K, Forni LG, Gomersall CD, Govil D, Honore PM, Joannes-Boyau O, Joannidis M, Korhonen AM, Lavrentieva A, Mehta RL, Palevsky P, Roessler E, Ronco C, Uchino S, Vazquez JA, Vidal Andrade E, Webb S, Kellum JA. Epidemiology of acute kidney injury in critically ill patients: the multinational AKI-EPI study. Intensive Care Med. 2015 Aug;41(8):1411-23. doi: 10.1007/s00134-015-3934-7. Epub 2015 Jul 11. PMID 26162677
- [Background] Vincent JL, Sakr Y, Sprung CL, Ranieri VM, Reinhart K, Gerlach H, Moreno R, Carlet J, Le Gall JR, Payen D; Sepsis Occurrence in Acutely Ill Patients Investigators. Sepsis in European intensive care units: results of the SOAP study. Crit Care Med. 2006 Feb;34(2):344-53. doi: 10.1097/01.ccm.0000194725.48928.3a. PMID 16424713
- [Background] Case J, Khan S, Khalid R, Khan A. Epidemiology of acute kidney injury in the intensive care unit. Crit Care Res Pract. 2013;2013:479730. doi: 10.1155/2013/479730. Epub 2013 Mar 21. PMID 23573420
- [Background] Chawla LS, Amdur RL, Amodeo S, Kimmel PL, Palant CE. The severity of acute kidney injury predicts progression to chronic kidney disease. Kidney Int. 2011 Jun;79(12):1361-9. doi: 10.1038/ki.2011.42. Epub 2011 Mar 23. PMID 21430640
- [Background] Zarjou A, Agarwal A. Sepsis and acute kidney injury. J Am Soc Nephrol. 2011 Jun;22(6):999-1006. doi: 10.1681/ASN.2010050484. Epub 2011 May 12. PMID 21566052
- [Background] Andreini C, Putignano V, Rosato A, Banci L. The human iron-proteome. Metallomics. 2018 Sep 19;10(9):1223-1231. doi: 10.1039/c8mt00146d. PMID 30095136
- [Background] Alnuwaysir RIS, Hoes MF, van Veldhuisen DJ, van der Meer P, Grote Beverborg N. Iron Deficiency in Heart Failure: Mechanisms and Pathophysiology. J Clin Med. 2021 Dec 27;11(1):125. doi: 10.3390/jcm11010125. PMID 35011874
- [Background] Melenovsky V, Petrak J, Mracek T, Benes J, Borlaug BA, Nuskova H, Pluhacek T, Spatenka J, Kovalcikova J, Drahota Z, Kautzner J, Pirk J, Houstek J. Myocardial iron content and mitochondrial function in human heart failure: a direct tissue analysis. Eur J Heart Fail. 2017 Apr;19(4):522-530. doi: 10.1002/ejhf.640. Epub 2016 Sep 19. PMID 27647766
- [Background] Hepokoski M, Singh P. Mitochondria as mediators of systemic inflammation and organ cross talk in acute kidney injury. Am J Physiol Renal Physiol. 2022 Jun 1;322(6):F589-F596. doi: 10.1152/ajprenal.00372.2021. Epub 2022 Apr 4. PMID 35379000

DOCUMENTS (1):
  • Study Protocol (2023-06-29): https://cdn.clinicaltrials.gov/large-docs/27/NCT05960227/Prot_000.pdf